CLINICAL TRIAL: NCT05052320
Title: Audiological Assessment of Recovered Covid 19 Subjects.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa kamal Mostafa Mohamed, Resident doctor, Assiut University
Other Study IDs: AARC19
Record Dates: First submitted 2021-09-17; First posted 2021-09-22 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Covid 19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Audiological assessment — TO assess audiological profile in recovered covid19 subjects

SUMMARY:
To assess the audiological profile in recovered covid 19 subjects in comparison with control group.

DETAILED DESCRIPTION:
The outbreak of novel Severe Acute Respiratory Syndrome Corona virus type 2 (nSARS-CoV-2) infection in Wuhan, China in December 2019 has had impact on the world, resulting in over 2.2 million deaths globally The world envisioned sufferings of high proportions of losses in terms of health,finances and importantly, life.

The common symptoms including fever, cough, fatigue and gastrointestinal disorders have been well documented. Sensorineural hearing loss has been more commonly implicated in these patients although a few have exhibited conductive hearing loss. theViral upper respiratory tract infections have linked to new cases of otitis media. Although There is some controversy regarding the significance of viral species, but the human corona virus has been isolated from middle ear fluid and linked to otitis media in children. Most patients affected are asymptomatic or experience mild symptoms.

Various theories explaining the involvement of the ear following covid infection have been pos tulated, which include immune mediated damage,haematogenous spread, ischaemia theory, inflammation of auditory pathway components, presence of angiotensin converting enzyme receptors (ACE2) receptors in neurons and glial cell.

The hearing loss in COVID-19 could also be the consequence of therapy with chloroquine and hydroxychloroquine, which are part of clinical practice guidelines for COVID-19 treatment in several countries . These drugs are used for the treatment of malaria and some chronic inflammatory diseases as well. It is well known that these medications can induce hearing loss. Ototoxicity of chloroquine and hydroxy- chloroquine is the result of inner ear damage . The recommended dose of these drugs for COVID-19 treatment is higher than for malaria; therefore, ototoxic effect could be higher.Though many vaccines were intro- duced, the disease has hit second and third waves in many countries, elevating the number of infected individuals getting infected .

Some studies reported that the COVID-19 group had significantly poorerhearing thresholds at high frequencies. In addition, the amplitudes of transient evoked otoacoustic emissions ,in two of thesestudies were significantly lower for the COVID-19 group.

ELIGIBILITY:
Inclusion Criteria:

* Age 18_50

Exclusion Criteria:

1. History of previous ear symptoms, tympanic membrane perforations,ear trauma or ear surgeries
2. Evidence of systemic illness as Diabetes mellitus, Renal disease, patients received ototoxic drugs.
3. Evidence of neurologicl or psychiatric disease.
4. covid 19 Patients not maintaining saturation and requiring O2 support and intensive care unit patient.

Ages: 18 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: Male or female subjects have recovered from covid 19 ..their age from 18_50
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Audiological assessment of recovered covid 19 subjects | base line
  To evaluate the audiological profile of recoveredcovid 19 subjects in comparison with control group

REFERENCES:
- [Background] Fancello V, Hatzopoulos S, Corazzi V, Bianchini C, Skarzynska MB, Pelucchi S, Skarzynski PH, Ciorba A. SARS-CoV-2 (COVID-19) and audio-vestibular disorders. Int J Immunopathol Pharmacol. 2021 Jan-Dec;35:20587384211027373. doi: 10.1177/20587384211027373. PMID 34142589
- [Result] Almufarrij I, Munro KJ. One year on: an updated systematic review of SARS-CoV-2, COVID-19 and audio-vestibular symptoms. Int J Audiol. 2021 Dec;60(12):935-945. doi: 10.1080/14992027.2021.1896793. Epub 2021 Mar 22. PMID 33750252
- [Result] Dharmarajan S, Bharathi MB, Sivapuram K, Prakash BG, Madhan S, Madhu A, Devi GN, Aliya SA, Ramya SB. Hearing Loss-a Camouflaged Manifestation of COVID 19 Infection. Indian J Otolaryngol Head Neck Surg. 2021 Dec;73(4):494-498. doi: 10.1007/s12070-021-02581-1. Epub 2021 May 10. PMID 33996529
- [Result] Dusan M, Milan S, Nikola D. COVID-19 caused hearing loss. Eur Arch Otorhinolaryngol. 2022 May;279(5):2363-2372. doi: 10.1007/s00405-021-06951-x. Epub 2021 Jul 8. PMID 34235578